NCT05305443 COVID-19 Treatment Cascade Optimization Study Protocol & Informed Consent 2/28/2023

# UNIVERSITY OF ILLINOIS URBANA-CHAMPAIGN

#### Office of the Vice Chancellor for Research & Innovation

Office for the Protection of Research Subjects 805 W. Pennsylvania Ave., MC-095 Urbana, IL 61801-4822

### **Notice of Approval: Continuing**

February 28, 2023

Principal Investigator Liliane Windsor CC Heather Perkins

Protocol Title COVID-19 Treatment Cascade Optimization Study

Protocol Number 22606

Funding Source National Institute of Health (NIH)

Review Type Full Board Status Active

Risk Determination More than minimal risk
Approval Date February 28, 2023
Expiration Date February 27, 2024

This letter authorizes the use of human subjects in the above protocol. The University of Illinois at Urbana-Champaign Institutional Review Board (IRB) has reviewed and approved the research study as described.

The Principal Investigator of this study is responsible for:

- Conducting research in a manner consistent with the requirements of the University and federal regulations found at 45 CFR 46.
- Using the approved consent documents, with the footer, from this approved package.
- · Requesting approval from the IRB prior to implementing modifications.
- Notifying OPRS of any problems involving human subjects, including unanticipated events, participant complaints, or protocol deviations.
- · Notifying OPRS of the completion of the study.



IRB Number: 22606

### **Human Subjects Research – Protocol Form**

### Guidelines for completing this research protocol:

- Please submit typed applications via email. Handwritten forms and hard copy forms will not be accepted.
- For items and questions that do not apply to the research, indicate as "not applicable."
- Provide information for all other items clearly and avoid using discipline specific jargon.
- Please only include text in the provided boxes. The text boxes will expand as they are typed in to accommodate large amounts of text.

### Before submitting this application, ensure that the following have been completed.

- Protocol Form is complete.
- Relevant CITI modules have been completed for all members of the research team at www.citiprogram.org.
- Informed consent/assent/parental permission document(s) are provided.
- Relevant waivers and appendices are provided.
- Recruitment materials are provided.
- Research materials (e.g. surveys, interview guides, etc.) are provided.
- Any relevant letters of support are provided.

Instructions on the non-exempt review process and guidance to submitting applications, can be found on the OPRS <u>website</u>. You may also contact OPRS by email at <u>irb@illinois.edu</u> or phone at 217-333-2670.

Submit completed applications via email to: irb@illinois.edu.



| PI. Other individuals may serve as PI | <mark>lanual</mark> allows assistant, asso<br>after obtaining approval fro | • | |
|---|---|---|---|
| Last Name: Windsor | First Name: Liliane | Degree( | s): PhD |
| Dept. or Unit: Social Work Office Address: 2113 | | | |
| Street Address: 1010 W. Nevada St. | City: Urbana | State: IL | Zip Code: |
| Phone: 217-300-1782 E-mail: lwindsor@illinois.edu | | | |
| Urbana-Champaign Campus Status:<br>Non-visiting member of (Mark One) [<br>(Student Investigators cannot serve as | | Professional/Staf | f |
| Training Required CITI Training, Date of Co Additional training, Date of Comp | | st 3 years), 11/08 | 3/2022 |
| ection 2. RESEARCH TEAM 2A. Are there other investigators eng | aged in the recearch? | | |
| Yes (include a Research Team Forr No | _ | | |
| 2B. If yes, are any of the researchers | | | |
| Yes No | not amiliated with illinois? | | |
| Yes No | not amiliated with illinois? | | |
| Yes No ection 3. PROTOCOL TITLE | | red to as COVID- | 19 IL Study) |
| Yes No PROTOCOL TITLE COVID-19 Treatment Cascade Optimiz | | red to as COVID- | 19 IL Study) |
| Yes No Rection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimize Rection 4. FUNDING SOURCE | | red to as COVID- | -19 IL Study) |
| Yes No PROTOCOL TITLE COVID-19 Treatment Cascade Optimize ection 4. FUNDING SOURCE | ation Study (Here after refe | | |
| Yes No ection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimize ection 4. FUNDING SOURCE 4A. Is the research funded? | ation Study (Here after refe | | |
| Yes No ection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimiz ection 4. FUNDING SOURCE 4A. Is the research funded? Research is not funded and is not Research is funded (funding decise) Funding decision is pending. Fund | ation Study (Here after refe<br>pending a funding decision<br>ion has been made).<br>ding proposal submission da | (Proceed to Secti | on 5). |
| Yes No ection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimiz ection 4. FUNDING SOURCE 4A. Is the research funded? Research is not funded and is not Research is funded (funding decis Funding decision is pending. Fundamental Fu | pending a funding decision ion has been made). | (Proceed to Secti<br>te: 07/07/2021- J | on 5). |
| Yes No ection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimiz ection 4. FUNDING SOURCE 4A. Is the research funded? Research is not funded and is not Research is funded (funding decis) Funding decision is pending. Fund 4B. Indicate the source of the funding University of Illinois Department, ( | pending a funding decision ion has been made). | (Proceed to Secti<br>te: 07/07/2021- J | on 5). |
| Yes No Rection 3. PROTOCOL TITLE COVID-19 Treatment Cascade Optimiz Rection 4. FUNDING SOURCE 4A. Is the research funded? Research is not funded and is not Research is funded (funding decision is pending. Fundamental Fu | pending a funding decision ion has been made). ding proposal submission data. College or Campus, please sp | (Proceed to Secti<br>te: 07/07/2021- J | on 5). |

<sup>&</sup>lt;sup>2</sup> Clarify whether or not the sponsor requires the protocol adhere to ICH GCP (E6) standards

| OFFICE FOR THE PROTECTION OF RESEARCH SUBJECTS | | UNIVERSITY OF ILLINOIS AT URBANA-CHAMPAIGN | | |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 02/07/2020 |

 $<sup>^{1}</sup>$  Clarify whether or not sponsor requires specific language in the contractual agreement that impacts human subjects research



## Office for the Protection of Research Subjects

### **Protocol Form**

| State of Illinois Department or Agency, <i>please specify</i> : |
|---|
| Other, please specify: |
| 4C. Sponsor-assigned grant number, if known: 1U01AI169469 - 01 |
| 4D. A complete copy of the funding proposal or contract is attached. |
| Attached, please specify title: COVID-19 Treatment Cascade Optimization Study |
| 4E. Funding Agency Official To Be Notified of IRB Approval (if Applicable) |
| Name: Program Officer TBD- Erin Khandjian, Grants Management Specialist |
| Agency: NIAID/NIH |
| E-mail: Erin.khandjian@nih.gov |
| <b>Phone:</b> 301-761-6557 |
| Section 5. CONFLICTS OF INTEREST |
| Please indicate below whether any investigators or members of their immediate families have any of |
| the following. If the answer to any of the following items is yes, please submit the University of Illinois |
| approved conflict management plan. If you have any questions about conflicts of interest, contact |
| coi@illinois.edu. |
| <b>5A.</b> Financial interest or fiduciary relationship with the research sponsor (e.g. investigator is a consultant |
| for the research sponsor). 🗌 Yes 🔀 No |
| <b>5B.</b> Financial interest or fiduciary relationship that is related to the research (e.g. investigator owns a |
| startup company, and the intellectual property developed in this protocol may be useful to the |
| company). 🗌 Yes 🔀 No |
| <b>5C.</b> Two or more members of the same family are acting as research team members on this protocol. |
| │ |

### Section 6. SUMMARY & PURPOSE OF RESEARCH

### 6A. In lay language, briefly summarize the objective and significance of the research.

COVID-19 has impacted the health and social fabric of individuals and families living across the United States; and it has disproportionately affected people living in urban communities with co-morbidities, those working in high-risk settings, refusing or unable to adhere to CDC guidelines, and more. Social determinants of health (SDH), such as stigma, racial discrimination, xenophobia, incarceration, and poverty have been associated with increased exposure to COVID-19 and increased deaths. Marginalized communities, defined as low-income and racial/ethnic minority neighborhoods, where residents experience increased barriers (e.g., inadequate housing, high-risk jobs) to prevention and treatment, bear disproportionately higher rates of co-morbidities associated with more severe cases of COVID-19. While effective and potent vaccines are becoming more available, it will take time to reach herd immunity and it is unclear how long newly-developed vaccines provide protection and how effective they are against emerging variants. Therefore, prevention methods recommended by the Centers for Disease Control and Prevention (CDC) – i.e., testing, hand-washing, social distancing, contact tracing, vaccination, and quarantine – are essential to reduce the rates of COVID-19 in marginalized



communities. Research about COVID-19 testing and vaccine uptake in these communities must occur in real time and it must account for the fast-changing landscape of the pandemic, including the impact of vaccine availability on testing uptake. Two cost-effective, evidence-based, and culturally appropriate interventions have been effective in engaging people in HIV prevention and treatment – these can be adapted and tested to help address COVID-19 prevention needs. Specifically, Navigation Services (NS) have been shown to increase HIV testing and adherence to treatment while addressing structural barriers that deter treatment engagement in high-risk communities; and Brief Counseling (BC) has been shown to increase HIV treatment engagement.

Dr. Windsor has an ongoing grant (3 R01 MD010629-04S2 – From here after referred to as COVID-19 NJ Study)) which aims to optimize an adaptive intervention to increase testing, and access to treatment and to prevention of COVID-19 infections in a medically or socially vulnerable sample of 670 people in Essex County, NJ. The COVID-19 NJ Study is under the North Jersey Community Research Initiative (NJCRI) IRB oversight, entitled *Optimization of a new adaptive intervention to increase COVID-19 testing among people at high risk in an urban community*, Protocol #: CWCOVIDSUPP-UIUC-NJCRI 102497-18274-267805 and has a reliance agreement in place with UIUC.

The new project, COVID-19 IL Study, which is being reviewed by the UIUC IRB, proposes to expand the NJ project to include a sample of 548 people in Illinois. We will use the same protocol that was used in NJ in addition to de-identified data that is currently being collected by the COVID-19 NJ Study. The final study sample will include 670 people from NJ and 548 people from IL for a total of 1,218. Data from the 670 people in NJ will be treated as secondary data and data from the 548 people in IL will be treated as primary data under the COVID-19 IL Study IRB protocol.

The COVID-19 IL Study will use Multiphase Optimization Strategy (MOST) and Community-Based Participatory Research (CBPR) principles and best practices to help facilitate recruitment and to make results readily available to the population. Illinois participants will be randomized two separate times: First, into two distinct groups to receive: (1) navigation services or (2) informational brochure. We aim to help participants to get a COVID-19 test between baseline and the first follow-up (7 days post baseline). Second, after completing the first follow-up, participants are then randomized again to continue with the original intervention or switch to a new one. We then collect data at 2; 5; 12; and 24 weeks post-baseline follow-ups.

The COVID-19 IL Study specific aims include:

Primary Aims: (1) To examine the effectiveness of an adaptive intervention to increase COVID-19 testing and adherence to CDC-recommendations of preventive behaviors – social distancing, hand-washing, mask-wearing, vaccination- on comparable but distinct samples. We will control for baseline, time, demographics and COVID risk; (2) To examine the immediate and medium-term impact of the adaptive intervention on COVID testing and adherence to recommendations by collecting follow up data at 2,5,12, and 24 weeks post baseline.



## Office for the Protection of Research Subjects

## **Protocol Form**

| Implementation aim: To collect intervention implementation data (context, cost, barriers, lessons learned) and develop implementation materials (facilitator training, intervention manual, treatment fidelity measure). |
|---|
| 6B. Indicate if your research includes any of the following: |
| Secondary data (use of data collected for purposes other than the current research project) Deidentified collected data by the COVID-19 NJ Study, described in final paragraph of 6A and COVID-19 |
| testing results collected from CBHC. |
| Data collected internationally (include International Research Form) |
| Translated documents (include <u>Certificate of Translation Form</u> and translated documents) |
| Research activities will take place at Carle (include documentation (email or letter) from Carle stating |
| that the review of your Research Services Request Form is complete) |
| 6C. Letters of support from outside institutions or entities that are allowing recruitment, research, or record access at their site(s) are attached. Yes Not Applicable |
| Letters of support from NJCRI and CBHC are in the NIH proposal (p.129- 132 of the attached proposal |
| PDF) |
| Section 7. PROCEDURES |
| 7A. Select all research methods and/or data sources that apply. |
| Surveys or questionnaires, select all that apply: Paper Telephone Online |
| Focus groups ("Critical Dialogue" Sessions) |
| Field work or ethnography |
| Standardized written, oral, or visual tests |
| Taste or smell testing |
| Intervention or experimental manipulation |
| Exercise and muscular strength testing |
| Noninvasive procedures to collect biological specimens (e.g., hair and nail clippings, saliva, etc.) |
| Noninvasive procedures to collect physiological data (e.g., physical sensors, electrocardiography, etc.) |
| Procedures involving radiation |
| Recording audio and/or video and/or taking photographs Recording other imaging |
| Materials that have already been collected or already exist, specify source of data: De-identified data |
| <del>-</del> |
| collected at another project that is led by the PI, Dr. Windsor in New Jersey at NJCRI using the same |
| <del>_</del> |



## Office for the Protection of Research Subjects

## **Protocol Form**

| | FERPA-protected data |
|---|---|
| | GDPR-protected data |
| | Other, please specify: |
| 7B | 3. List all testing instruments, surveys, interview guides, etc. that will be used in this research. |
| Eli | Eligibility Screener Enrollment |
| Ва | Baseline Survey |
| Fo | Follow up 1 to 4 Survey |
| Br | ochures |
| Dr | rafts or final copies of all research materials are attached. 🔀 Yes |
| 70 | C. List approximate study dates. 03/10/2022- 12/31/2023 |
| 70 | D. What is the duration of participants' involvement? 6 months |
| <b>7</b> E | . How many times will participants engage in research activities? Participation will complete 1 |
| ba | seline and 4 follow up assessments. Those randomized to Navigation Services will complete at least |
| or | ne phone session of up to 30 minutes on the phone. They may request as many navigation sessions as |
| th | ey need. Those randomized to Brief Counseling will complete one 15 minutes long phone session. |
| Th | nose randomized to Critical Dialogue will complete one 60 minutes long session in-person or online. |
| | . Narratively describe the research procedures in the order in which they will be conducted. |
| | is study will track participants for six months in order to capture changes over time in COVID-19 |
| | sting and adherence to public health recommendations. We will use a Sequential, Multiple Assignment |
| | andomized Trial (SMART) with a total sample of 1,218 COVID-19 medically and socially vulnerable |
| - | eople, 548 of which will be primary data collection and 670 will be secondary data. All participants will |
| | ceive at least one intervention and no more than two interventions, depending upon randomization. |
| | ter having been determined eligible through a brief phone screening process, participants will be |
| in | vited to provide consent to participate and complete the baseline online. Those interested in the study |
| wi | ill call the study phone. A research assistant or outreach worker will complete the phone screening |
| wi | th the participant to determine eligibility. If eligible, they will be asked to provide alternative forms of |
| со | ntact in case we are unable to reach them. The staff will explain that they will let the alternative |
| со | ntact know we are looking for the participant because it is time for them to complete their follow-up |
| su | rvey. Participants may choose not to provide any contacts. Those who complete the baseline will then |
| be | e randomized by Redcap to either receive Navigation Services or Brochure: |
| Na | avigation Services (NS): Navigation services include assessment and support with service referrals. Each |
| | articipant randomized to this intervention will meet with a peer navigator in person or on Zoom |
| - | onferencing for 30 minutes to go over results from their social and health needs assessment that is |
| | trieved from the base-line survey. The navigator shares information about COVID-19, answers |
| | uestions about testing, and makes referrals to other needed services (e.g., housing, food, mental |
| | ealth, employment, transportation, primary care). The participant is then referred to the testing site |
| | nd encouraged to get tested as soon as possible. The peer navigator calls participants who consent to |

follow up, find out what services they received, and what services they still need. The frequency of sessions is decided between the participant and the navigator. The peer navigator can then make new



referrals and help participants address identified barriers to services. All referrals and referral outcomes will be tracked and entered into the project database.

<u>Brochure:</u> This intervention includes two different electronic brochures: One with information about COVID-19 testing (including where and how to get tested), and one with information about COVID-19 prevention and treatment. The brochures will be updated in real time to reflect the most recent CDC public health recommendations. Brochures will be e-mailed to all participants automatically by Redcap upon randomization and one week after they complete the baseline.

Once randomized, all participants will receive the brochure that includes information about testing at CBHC. Navigators will speak to their clients about testing, and, if the participant is interested, they can schedule the COVID-19 test for participants. Note participants will not be pressured to test. They will simply receive the information on how to do so and we will ask them to do it prior to completing their follow-up, if they choose to get tested. Home tests will not be accepted for the purposes of the study.

One week post-baseline, participants will complete the first follow-up survey. Those who received a COVID-19 test between baseline and Follow-up 1 will be randomized to either continue to receive their original intervention (NS or Brochure) or to switch to receive Brief Counseling. Those who fail to get a COVID-19 test between baseline and first follow-up will be randomized to continue the original intervention (NS or Brochure) or switch to receive Critical Dialogue:

<u>Brief Counseling (BC):</u> Brief Counseling is a 15-minute post-COVID-19 test session delivered by a trained licensed clinician in person or via Zoom Conferencing. In the session, the clinician shares the test results and offers recommendations and information about COVID-19 treatment and prevention. Clinicians will be members of the research team and employed by CBHC.

<u>Critical Dialogue (CD):</u> Critical Dialogue includes one two-hour "focus group" session facilitated in person or online by a trained licensed facilitator. Group critical dialogue is prompted by thematic images developed by the Newark Community Collaborative Board (NCCB) to foster a deeper understanding of how systematic stigma, feelings of rage as victims of discrimination, and/or apathy may impact participants' beliefs and behaviors related to COVID-19 and empower participants to make critical choices to protect their health and the health of their communities.

COVID-19 test procedures and HIPPA protected data collection and sharing: Enrolled participants interested in getting tested for COVID-19 will either come into CBHC or meet the trained outreach worker to collect the sample. CBHC holds a Clinical Laboratory Improvement Amendment (CLIA) Certificate of Waiver and uses the Lumira Dx SARS-CoV-2 Ag Test (see attached instruction manual). The outreach worker will be using N-95 mask and gloves. Participants are asked to collect their own nasal sample and hand it over to the outreach worker who processes it. It takes 15 minutes to obtain the test results and participants are informed immediately. They receive the study brochure that provides



information about how to prevent COVID-19 and what to do if tested positive. As soon as the results come out, the outreach worker logs into Redcap and records the test completion date and results.

In cases where the sample is collected outside of CBHC, the participant will be asked to collect the sample following the instructions, place it into a plastic bag, and hand it to the outreach worker. The collection bag will have the participants' study code number written on it and it is transported in a cooler container back to CBHC. Once the sample is processed, the outreach worker calls the participant to provide the test results and logs the information in Redcap. They receive the brochure when they turn in the sample.

With participants' permission, we will share the COVID-19 test results and some identifying information (e.g., zip codes) with the Duke Clinical Research Institute (DCRI). HIPPA data will be downloaded from Redcap automatically including only data that was authorized by participants to be shared with the CDCC. This will be a CVS file which is downloaded into Box Health. The file is then uploaded weekly into the Duke data portal (see attached CDCC Data guidance pdf).

Participants who report not getting tested in follow-up 3 will be invited to participate in a Critical Dialogue session before completing Follow-up 4.

All participants will be asked to complete follow ups 4 and 5. We will collect screening data via phone, and in-person baseline assessment, and follow- ups at 2, 5, 12 and 24 weeks follow-ups. Participants will be encouraged to complete the surveys online, using their phones, a tablet, or computer. They can also request to meet the outreach workers at CBHC or a public place to complete the data collection using a study tablet, as long as they agree to adhere to the most current public health recommendations (e.g., social distancing).

After each assessment, participants will be asked to provide extensive locator information, on forms used for the parent study, including formal and informal contacts who can reach the participant in a variety of contingencies. During the follow-up period, outreach workers will maintain monthly contact with participants by mail or phone and will update locator information. Randomization and data collection will be done online using Redcap. We will voice record all Critical Dialogue sessions with participants' consent and will randomly select 20% of them for analysis.

The research team will randomly select 35 participants at each site who decline to be tested for COVID-19 and invite each of them to complete an in-depth, one-on-one, qualitative interview lasting about 30 minutes. After providing written informed consent, participants will be assigned code names and asked to talk about their experiences with the intervention, barriers they faced to testing and adhering to public health guidelines, and their ideas about how to address these barriers. The interviews will be digitally voice-recorded, transcribed and entered into Atlas.ti for storage and analysis. Transcripts and Atlas.ti files will be identified only by code name.



Additionally, data from the COVID-19 NJ Study will be analyzed. These data include the exact same surveys as the data being collected in Illinois. The data is being collected under NJCRI's IRB number. UIUC deferred to the NJCRI IRB because all the NJ data is being collected there. The NJ data will be deidentified and shared electronically by the NJ research assistant using Box. The NJ data will then be merged with the Illinois data for analysis.

## The figure below illustrates the study design: 1<sup>st</sup> stage intervention



COVID- 19 Testing

### Section 8. PERFORMANCE SITES TO INCLUDE INTERNATIONAL, SCHOOL, AND COLLABORATIVE **STUDIES**

8A. List all research sites for the protocol. For non-University of Illinois at Urbana-Champaign sites, describe their status of approval and provide contact information for the site. If the site has an IRB, note whether the IRB has approved the research or plans to defer review to the University of Illinois at Urbana-Champaign.

### **Performances Sites** Comprehensive Behavioral Health Center (CBHC)- East St. Louis, IL Joe Harper, Executive Director (618) 482-7330 jharper@cbhc1.org CBHC will defer to UIUC IRB

North Jersey Community Research Initiative (NJCRI), Newark, NJ FWA00001870



## Office for the Protection of Research Subjects

## **Protocol Form**

| | James Oleske, MD, MPH Chairman of the NJCRI IRB |
|---|---|
| | oleskejm@njms.rutgers.edu |
| | Corey DeStefano, Director of Research |
| | c.rosmarin@njcri.org |
| | (973) 483-3444 |
| | NJCRI will defer to UIUC IRB |
| #3 | University of Michigan (UM) FWA00004969 |
| "3 | Mary Donnelly, Single IRB Coordinator, mardonne@umich.edu |
| | Office: (734) 936-0933, irbhsbs@umich.edu |
| | UM will defer to UIUC IRB |
| If th | ere are additional performance sites, include them on an attachment and check here: |
| | Is this a multi-center study in which the Illinois investigator is the lead investigator, or the |
| | versity of Illinois at Urbana-Champaign is the lead site? X Yes No |
| | es, answer 8C and 8D. If no, proceed to Section 8E. |
| | Who is the prime recipient of funding, if funded? UIUC |
| | What is the management and communication plan for information that might be relevant to the |
| - | ection of research subjects (e.g. unanticipated problems involving risks to subjects, interim results, |
| | protocol modifications)? Dr. Windsor and Mr. Harper will be responsible for overseeing all data |
| | ection and processing. While the proposed study does not seek to test the effectiveness of drugs or a |
| | lical device delivered in multiple sites, it will test an adaptive intervention in communities with |
| | ginalized populations and there is potential for harm. Thus, we developed a Data and Safety |
| | nitoring Plan (DSMP) and will create an independent Data Safety and Monitoring Board (DSMB) |
| | uding clinical, intervention, community members, and statistical experts, to conduct periodic |
| inde | pendent analyses of the evaluation data in the data collection phase. |
| | research staff member who learns of an adverse event is responsible for reporting the event to the |
| | cipal Investigators (PI), who are in turn responsible for discussing the event to make a joint decision |
| | ut whether the event is serious or non-serious. Events will be categorized as adverse or serious |
| | erse according to NIH guidelines: "Adverse events (AEs) are defined as any untoward medical |
| | urrence that may present itself during treatment or administration of an intervention, and which may |
| | nay not have a causal relationship with the treatment. Serious adverse events (SAEs) are defined as |
| • | medical occurrence that results in death; is life-threatening; requires inpatient hospitalization or |
| - | ongation of existing hospitalization; creates persistent or significant disability/incapacity, or a |
| | genital anomaly/birth defects." As such, adverse events (AEs) occurring during the course of the |
| | y will be collected, documented, and reported to the PIs. Each week a study investigator will review |
| the | AE Forms from the previous week for events that were reported as new or continuing. |
| ۸ ۵۰۰ | CAE will be reported to the IDD within 40 hours of the accurrence. The report of CAEs will include |
| • | SAE will be reported to the IRB within 48 hours of the occurrence. The report of SAEs will include |
| | ther they were expected or unexpected, a rating of severity of the event, a brief narrative summary |
| of th | ne event, a determination of whether a causal relationship existed between the study procedures |



| and the event, whether the informed consent should be changed as a result of the event and whether all enrolled participants should be notified of the event. Finally, as part of the annual progress report (noncompeting continuation application) to NIH, we would provide summary information on all SAEs |
|---|
| that have occurred during that year. |
| Any actions taken by the IRB will be reported promptly to NIH via the Project Officer or appropriate parties. |
| Additionally, the PIs and Dr. Sarol will closely monitor the validity and integrity of the data on an ongoing basis. The DSMB with also conduct biannual monitoring of the data through spot checks and |
| independent preliminary analysis of the data. For instance, the PIs and the project staff will meet |
| regularly with project interviewers to review assessments and coding of incoming data. The PIs will be |
| responsible for ensuring that data are being coded, entered and cleaned appropriately. The full research |
| team will meet every week for 120 minutes to review all aspects of the research study. |
| 8E. If subjects will be recruited from Illinois public or private elementary or secondary schools, |
| additional deadlines and procedures may apply. Criminal background clearances might be required. |
| Special consideration must be given to the exclusion of protected populations. Please contact the |
| <u>School University Research Relations</u> ( <u>researchplacements@education.illinois.edu</u> ) for more |
| information. Select one: Illinois schools will be used Illinois schools will not be used |

### Section 9. SUBJECT ENROLLMENT GOAL & EQUITABLE SELECTION OF SUBJECTS

| 9A. For each performance site, indicate the estimated total number of participants. | | | | |
|---|---|---|---|---|
| Perf | formance Site | # Male | # Female | Total |
| #1 | СВНС | 252 | 295 | 548 |
| #2 | NJCRI (oversight by NJCRI IRB) | 328 | 341 | 670 |
| #3 | UM | 0 | 0 | 0 |
| TOT | ALS | 580 | 636 | 1218 |
| If a | dditional performance sites are included on an af | ttachment, check l | here: | |
| 9B. | Select all participant populations that will be red | cruited. | | |
| Age | Age: | | | |
| $\boxtimes$ | Adults (18+ years old) | | | |
| Minors (≤17 years old) | | | | |
| Specific age range, <i>please specify</i> : | | | | |
| Gender: | | | | |
| No targeted gender (both men and women will be recruited/included) | | | | |
| | Targeted gender, <i>please indicate</i> : 🔲 Men/boys 🛚 | ☐ Women/girls ☐ | ] Other, <i>please sp</i> | ecify: |
| Rac | e/Ethnicity: | | | |
| No targeted race or ethnicity (all races and ethnicities will be recruited/included) | | | | |
| | Targeted race or ethnicity, please specify: | | | |



## Office for the Protection of Research Subjects

## **Protocol Form**

| College Students: |
|---|
| No targeted college population |
| UIUC general student body |
| Targeted UIUC student population, provide the instructor or course information, name of the |
| departmental subject pool, or other specific characteristics: |
| Students at institution(s) other than UIUC, please specify: |
| Any research with students on UIUC's campus needs to be registered with the Office of the Dean of |
| <u>Students</u> . |
| Other: |
| ☐ Inpatients |
| Outpatients |
| People who are illiterate or educationally disadvantaged |
| People who are low-income or economically disadvantaged |
| People with mental or cognitive disabilities or otherwise impaired decision-making capacities |
| Adults with legal guardians |
| People who are non-English speaking |
| People with physical disabilities |
| Pregnant or lactating women, human fetuses, and/or neonates |
| Prisoners or people with otherwise limited civil freedoms |
| Other, please specify: target population faces disproportionate COVID-19 risks due to employment as |
| essential workers, poverty, inadequate or unstable housing, and underlying medical conditions. |
| 9C. Describe additional safeguards included in the protocol to protect the rights and welfare of the |
| populations selected above. |
| To avoid possible violations of confidentiality, project staff are trained to carefully follow detailed |
| procedures designed to assure that no information about any participant (or others they may mention) |
| will be given to law enforcement, other government agencies, or anyone but research staff. Every |
| member of the research team and all members of the NCCB and the Illinois Community Collaborative |
| Board (ICCB) will be required to undergo human subject protection training and provide a certificate of |
| completion to the |
| IRB prior to any contact with human subjects. Standards of confidentiality include the use of code |
| numbers and code names for participants and other individuals they may mention. The only place |
| participants' names or other identifying information will appear is on informed consent forms and |
| locator forms (used for follow-up interviews after the baseline). These forms will be kept electronically in |
| REDCAP, in a folder separate from the data. Only full time, trained staff in the project including the |
| outreach works, project coordinator, research assistant, and PIs will have access to these files. Peer |
| navigators will not have access to data from the individuals that are randomized into their groups. They |
| will receive a report from RedCAP highlighting any reported risk for COVID-19 exposure that they will be |
| discussing with the participant during the navigation. |
| The electronic files generated through data collection will be identified by code numbers and |



codenames only and kept in password-protected devices/servers, separate from identifying information and available only to project staff. This helps to ensure that no identifying information will be disclosed in the unlikely event that computerized data are stolen or otherwise seen by unauthorized persons.) All identifying electronic data will be destroyed immediately after data analysis is completed. Signed consent forms will be kept for 3 years after study completion. Deidentified electronic data will be kept indefinitely. Participants may ask at any time to have recordings of their interview destroyed by calling/e-mailing one of the Principal Investigators at the numbers provided in the informed consent forms. Voice recordings will be kept indefinitely for data analysis. However, if we have reason to believe that any of these recordings contain information that can put any of our participants in danger of being harmed, we will destroy the recording.

Our interviewers are trained to watch participants carefully and will stop questioning if an individual appears uneasy. At every interview, participants will be informed that they may ask the interviewer to stop if they are feeling uncomfortable. Referrals to counselors are available if participants wish and trained clinical counselors are available at CHBC in the event that someone may need immediate assistance, whether it is during data collection or during the intervention sessions. Dr. Windsor, Dr. Benoit, and Mr. Harper will be available by phone at all times in case an emergency occurs. Clinical emergencies will be handled by treatment teams of experienced staff at CBCH under the leadership of Mr. Harper. Appropriate assessments will be conducted; treatment options will be recommended and followed through as necessary. CBHC routinely provides services to individuals with mental health and substance use disorders is fully equipped to address any potential emergencies either themselves or via referrals.

Finally, the research team and the clinical team will engage in weekly project meetings to discuss the progress of the study and identify, discuss, and address any potential issues.

### Section 10. INCLUSION/EXCLUSION

10A. List specific criteria for inclusion and exclusion of subjects in the study, including treatment and control groups.

Criteria for inclusion include:

- 18 years of age or older
- having high risk to contract COVID-19 or develop related complications
- able to Speak English at the 7<sup>th</sup> grade level
- able and willing to provide informed consent

10B. Explain how the inclusion/exclusion criteria will be assessed and by whom. If special expertise is required to evaluate screening responses or data, list who will make this evaluation and describe their training and experience.

A trained outreach worker will conduct a brief phone screening using the attached brief phone screening to obtain self-reported eligibility information including risk for contracting COVID-19 and developing related complications.



| <b>10C. Drafts or final copies of all screening materials are attached.</b> ⊠ Yes ☐ Not Applicable |
|---|
| 10D. Describe procedures to assure equitable selection of subjects. Justify the use of the groups |
| marked in Section 9B. Selection criteria that target one sex, race, or ethnic group require a clear |
| scientific rationale. |
| The proposed study does not include children because the adaptive intervention will focus on adult |
| behaviors and it would not be appropriate to include children. The staff has been trained to work with |
| adults and the parent grant only included individuals over the age of 18. Finally, the supplement includes |
| several interview questions regarding social determinants of health that children would not be able to |
| answer. Recruitment will be open to residents of both Essex County, NJ and St. Clair County, IL, but given |
| the location of the study sites, we expect that the vast majority of participants will come from the |
| Newark, NJ and East St. Louis, IL areas. As such, we estimate that our sample will approximate the |
| demographics of Newark and East St. Louis in terms of sex/gender, race and ethnicity. Because of this, |
| we anticipate that Black participants will be overrepresented in our sample. |
| Section 11. RECRUITMENT |
| 11A. Select all recruitment procedures that will be used. |
| Student subject pool, <i>please specify</i> : |
| Email distribution |
| MTurk, Qualtrics Panel, or similar online population, <i>please specify</i> : |
| US Mail |
| Flyers/brochures |
| Website ad, online announcement (e.g. eWeek), or other online recruitment, please specify: |
| Newspaper ad |
| Verbal announcement |
| Other, please specify: Street outreach |
| Not applicable (secondary data only) |
| 11B. Drafts or final copies of all recruitment materials (including verbal scripts) are attached. |
| Yes Not Applicable |
| 11C. For each group of participants, describe the details of the recruitment process. |
| We will enroll a sample of 548 in St. Clair County. The ICCB and outreach staff will post fliers at bus stops, |
| health care agencies, churches, bulletin boards, and social service agencies, giving consideration to the |
| demographic characteristics of those agencies' clients and of neighborhoods. Individual service providers |
| and potential participants will be asked to share the study's fliers in their neighborhoods, churches and |
| other meeting places. Those who are interested will call the study phone number that is listed on the |
| flyer. Street outreach will be used following social distancing protocol. All consenting CBHC clients will be |
| screened and those eligible will be invited to participate in the study. People interested in participating |
| will call the study's cell phone number. A trained outreach worker will conduct a brief phone screening |
| using the same brief phone screening that is currently being used in the Essex County, NJ to obtain self- |



| reported eligibility information including risk for contracting COVID-19 and developing related |
|---|
| complications. |
| Section 12. REMUNERATION AND PLAN FOR DISTRIBUTION |
| Refer to the University <u>Business and Financial Policies and Procedures</u> for further guidance on the |
| compensation process and reporting requirements. |
| 12A. Will subjects receive inducements or rewards before, during, or after participation? |
| ∑ Yes |
| If yes, complete the rest of Section 12. If no, proceed to Section 13. |
| 12B. Select all forms of remuneration that apply. |
| Cash, please specify amount: \$30 for baseline, \$40 per follow up, \$30 for group session, and \$50 for |
| the exit interview for a maximum possible of \$270 per individual |
| Check, please specify amount: |
| Gift Certificate, please specify amount: |
| Lottery, please specify amount: and odds: |
| Course Credit, please specify amount: and specify equivalent alternative activity: |
| Other, please specify: |
| 12C. Will payment be prorated before, during, or after participation? |
| Yes, please specify how: Payments will be received after completion of each survey during the study. |
| No |
| 12D. For each group of participants, describe the details of the remuneration plan, including how, |
| when and by whom they will be notified. |
| Participants will receive modest cash incentives for taking part in data collection activities. Each |
| participant will receive \$30 for completing the baseline assessment. Each participant will receive \$40 per |
| each of the four "follow up" visits. Each participant will receive \$30 for attending a one hour Critical |
| Dialogue session. The maximum amount possible for participation is \$270 per individual. |
| 12E. The information listed above is provided on the relevant consent forms. |
| ∑ Yes |

### **Section 13. RISKS & BENEFITS**

13A. Describe all known risks to the participants for the activities proposed, such as risks to the participants' physical well-being, privacy, dignity, self-respect, psyche, emotions, reputation, employability, and criminal and legal status. Risks must be described on consent forms.

The main potential risks of this study include inadvertent violation of confidentiality and emotional distress on the part of participants. The use of code names and numbers along with other procedures described below are intended to prevent violations of confidentiality. It is important to be aware that the prospect of testing positive for COVID-19 may be a cause of substantial fear and anxiety among



participants. We anticipate that more than half of our participants will be African American or Hispanic and may lack trust in medical science and practice as a legacy of medical mistreatment. Many participants will have lost loved ones to COVID-19 and all of them will be medically or socially vulnerable to poor outcomes if they become infected themselves. They live with disproportionate risk caused by any of several factors, including but not limited to employment as essential workers, poverty, inadequate or unstable housing and underlying medical conditions. CBHC has been operating as a primary provider of services in East St. Louis, IL for 50 years. It is, in general, a trusted source of care and services, but the COVID-19 pandemic is a recent, evolving development and much remains unknown about community perceptions.

It is also possible that participants who decline testing and attend Critical Dialogue sessions may be disturbed by sensitive questions raised during those sessions. Questions and discussions regarding stigma, racism, discrimination and structural inequality may cause anxiety, anger, suspicion, or other emotions. While we expect our sample to be predominantly African American, there will be some White and Latino participants as well and talking about racism in the group will elicit strong emotions. Differences among group members have the potential to harm or cause discomfort for a participant or to revive psychological dynamics that could threaten to renew old conflicts.

13B. Describe the steps that will be taken to minimize the risks listed above.

To avoid possible violations of confidentiality, project staff are trained to carefully follow detailed procedures designed to assure that no information about any participant (or others they may mention) will be given to anyone other than members of the research staff included in the IRB protocol. Every member of the research team and all NCCB and ICCB members will be required to undergo human subject protection training and provide a certificate of completion to the IRB prior to any contact with human participants. Standards of confidentiality include the use of code numbers and code names for participants and other individuals they may mention. The only place participants' names or other identifying information will appear is on informed consent forms and locator forms that are password protected in RedCap, the software used in the study. This identifying information is used for follow-up interviews after the baseline, to remind participants of Critical Dialogue group sessions if they are randomized to that condition and to locate participants if we are unable to reach them. Consent forms will be stored in locked filing cabinets at CBHC, separate from any data. Mr. Harper, the Project Principal Investigator at CBHC, will retain the keys to the filing cabinets at each location. Only outreach staff, Dr. Windsor, Mr. Harper, and the group facilitators will have access to the identifying information.

The electronic files generated through data collection will be identified by code numbers only and kept in password-protected and HIPAA-compliant devices/cloud, separate from identifying information and available only to project staff. This helps to ensure that no identifying information will be disclosed in the unlikely event that computerized data are stolen or otherwise seen by unauthorized persons. All identifying electronic data will be destroyed immediately after data collection is completed. Signed consent forms and audio recordings will be kept for 3 years after study completion. De-identified



electronic data will be kept indefinitely. Study participants may ask at any time to have recordings of their interview destroyed by calling/e-mailing one of the Principal Investigators at the numbers provided in the informed consent forms.

Participants will be protected by a Certificate of Confidentiality issued by the NIH. NIH issues COCs automatically upon funding approval. Under terms of the Certificate, the researchers cannot be forced to disclose information that may identify a participant, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. However, the Certificate cannot be used to resist a demand from United States Government personnel for information that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). Researchers may also disclose the identity of participants who report intentions to harm themselves or others or if researchers have knowledge those participants are abusing children or elderly persons

Our interviewers are trained to watch participants carefully and will stop questioning if an individual appears uneasy. At every interview, participants will be informed that they may ask the interviewer to stop if they are feeling uncomfortable. Referrals to counselors are available if participants wish and trained clinical counselors are available at CBHC in the event that someone may need immediate assistance, whether it is during data collection or during the intervention sessions. The Critical Dialogue is an intervention developed by Dr. Windsor and the NCCB, to ensure that the group discussions happen in a safe way, where everyone is encouraged to challenge their own assumptions by analyzing the evidence they have that supports or challenges their positions. This starts with operational components where the intervention is clearly described so that people know what to expect, and ground rules are collaboratively created and enforced during group discussions. In preliminary research on the intervention, there were many instances where the critical questions posed led to a heated dialogue where people were able to express their conflicting views while respecting each other and considering the possibility of changing their points of view. Dr. Windsor will train a doctoral level social work research assistant to facilitate the groups. The RA has a great deal of experience facilitating groups dealing with these sensitive topics and with this marginalized population. In the unlikely event a discussion escalates to the point that it may challenge the safety of the group, there is an emergency protocol in place where trained clinical staff and security can intervene and deflect potential violence or stabilize medical emergencies. During the development and testing stages of the intervention, with close to 700 participants, no adverse events occurred as a result of critical dialogue participation.

The IRBs of the collaborating institutions, the NJCRI, CBHC, and the University of Michigan, will defer oversight to the UIUC IRB. As the applicant agency, the University of Illinois Urbana-Champaign will ensure that all institutions adhere to IRB monitoring and will keep annual certificates from each institution on file. UIUC will execute an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Authorization Agreement with all other agencies. The Officials signing this Agreement will thereby



agree that their institutions may rely on the IRB of UIUC as the designated IRB for review and continuing oversight of its human subjects research described for this project. Dr. Windsor, Dr. Benoit, Mr. Harper, and Dr. Pinto will be available by phone at all times in case an emergency occurs. Any adverse event will be reported to the IRB and funding agency within 24 hours. Through our ICCB collaboration, we have excellent relationships with the community, including community members and agencies that we can mobilize in case the need arises (e.g., access to detox and emergency services, legal support clinics). Finally, the research team and the clinical team will engage in weekly project meetings to receive ongoing training, discuss the progress of the study and identify and address any potential issues. 13C. Indicate the risk level. No more than minimal risk (The probability and magnitude of harm or discomfort anticipated for participation in the proposed research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests). More than minimal risk (answer 13D) 13D. If you checked that the research is more than minimal risk, describe the provisions for monitoring the data to ensure the safety of subjects, such as who will monitor data and how often, what criteria will be used to stop the research, etc. The MPIs will oversee data management, including data storage, security, random assignment and quality assurance procedures, REDCap, software and hardware, and will ensure that all staff adheres to Human Subjects guidelines. Data management activities and procedures, including data confidentiality, will employ an electronic data management system to enhance efficiency, security and integrity of study data. The ICCB will also be updated during meetings on data management and adherence to IRB protocol. Additionally, integrity assessments will be conducted, which include: (1) a checklist completed by facilitators at the end of each intervention session to list the activities discussed in each session and participant attendance; (2) exit interview. The NCCB and ICCB will review preliminary findings presented by the MPIs on a bi-monthly basis to address any potential adverse reactions that may occur and any safety concerns that may arise. If any participants are found to be unresponsive to the intervention during the course of the study, the Board will discuss the case and the participant may be terminated from the study and referred to relevant services in the community. The MPIs will meet bi-weekly with study staff to review study protocol adherence and address any potential problems. MPI Windsor will have weekly supervision meetings with intervention facilitators to review results from fidelity ratings and address any potential deviance from intervention protocols.



### 13E. Describe the expected benefits of the research to the subjects and/or to society.

The potential benefits to participants in this study and other members of the community are significant and may be long lasting. Significant short-term benefits include detecting and treating cases of COVID-19 and preventing further transmission of the disease. While participants are enrolled in the study, referrals to resources to address social determinants of health (e.g., housing, food insecurity) may provide immediate tangible benefits. In addition, if participants express a need for mental health assistance at any time, the project team and the ICCB are well equipped to either provide service or make appropriate referrals. After engaging in the interventions, participants may experience increased feelings of empowerment and self-esteem, both of which have been associated with improved health outcomes. If the study succeeds in reducing medical mistrust and increasing health literacy, those benefits may belong-lasting. Both the short-term and long-term potential benefits of this study justify the potential risks involved in participation.

13F. Weigh the risks with regard to the benefits. Provide evidence that benefits outweigh risks.

Knowledge to be gained from this investigation is important for understanding and addressing COVID-19 morbidity and mortality disparities and potential barriers to testing among medically and socially vulnerable populations. The opportunity to engage residents of East St. Louis, IL in the proposed adaptive interventions is an opportunity to increase health literacy and reduce medical mistrust among a severely underserved population. This is vitally important in light of the contradictory and constantly changing information about COVID-19 being disseminated by federal and state governments and mass media. Moreover, because the knowledge generated by this study will be shared with other members of the RADx-UP consortium, it has the potential to improve access to prevention strategies, testing and treatment in vulnerable communities across the country. The value of the knowledge to be gained far outweigh the potential risks of participation described above, particularly when considering the precautions we have taken to minimize these risks. Although participants' risk of experiencing COVID-19 related distress is real, involvement in the study can also reduce fear and anxiety. As explained earlier, project staff will employ every effort to maintain confidentiality and to minimize any other potential risks; should a serious adverse event occur, it will be reported to the DSMB, Project Officer, funding agencies and the UIUC IRB within 48 hours. Adverse events will be tracked in a database and reviewed at each DSMB meeting. Our CBPR research to date indicates that community members themselves will be committed to assisting us in the successful and safe implementation of this project.

### Section 14. INFORMED CONSENT PROCESS TO INCLUDE: WAIVERS, ASSENTS, ALTERATIONS, ETC.

| 14A. Indicate all that apply for the consent/assent/parental permission process. |
|---|
| Written informed consent (assent) with a document signed by |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| Waiver of Documentation (signature) of Informed Consent (include the relevant Waiver Form) |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| Waiver of Informed Consent (include the relevant Waiver Form) |
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |



## Office for the Protection of Research Subjects

## **Protocol Form**

| Alteration of Informed Consent (include the relevant Alteration Form) |
|---|
| adult subjects parent(s) or guardian(s) adolescents aged 8–17 years |
| 14B. List all researchers who will obtain consent/assent/parental permission from participants. |
| Researchers who may participate in obtaining consent include the PIs (Windsor & Harper), |
| project coordinator, study outreach workers and research assistants at CBHC that will be trained |
| and approved as members of the research team by the UIUC IRB. Note we have not yet hired |
| the project coordinator nor the peer navigators. Staff will be added to the protocol as they are |
| hired and complete their IRB training. Only staff that have been approved by the IRB will have |
| contact with study participants. |
| <b>14C.</b> Describe the method for obtaining consent/assent/parental permission. Eligible individuals will |
| provide written informed consent before participating in the study. During the informed |
| consent process, the study outreach worker or research assistant will explain the study design in |
| detail, including its purpose, the source of funding, why individuals are invited to participate, |
| what they will be asked to do, how long the study will last and how many people are expected |
| to take part in the study. They will explain the processes of SARS antigen testing at CBHC and |
| randomization, the interventions being tested, potential sources of risk and discomfort and |
| measures designed to minimize both. They will answer all participant questions and will ask |
| participants to describe in their own words what they expect to do in the study before obtaining |
| signatures. Participants who do not comprehend the study description will not be enrolled. |
| Participants who would like some time to think before deciding will be able to take informed |
| consent material home with them for review and consideration. All participants who provide |
| written consent will receive a copy of the consent document which, in addition to the study |
| description outlined above, includes names and contact information (phone numbers and email) |
| for the Principal Investigators and for the appropriate ethics officials at the University of Illinois |
| Urbana-Champaign, the grantee institution. |
| 14D. Describe when consent/assent/parental permission will be obtained. Consent will be obtained |
| through a RedCAP survey that participants can complete online or at CBHC. |
| 14E. Will participants receive a copy of the consent form for their records? |
| Yes No, if no, explain: |
| 14F. Indicate factors that may interfere or influence the collection of voluntary informed |
| consent/assent/parental permission. |
| No known factors |
| Research will involve students enrolled in a course or program taught by a member of the research |
| team |
| Research will involve employees whose supervisor(s) is/are recruiting participants |
| Participants have a close relationship to the research team |



## Office for the Protection of Research Subjects

## **Protocol Form**

| Other, specify any relationship that exists between the research team and participants: |
|---|
| If applicable, describe the procedures to mitigate the above factors. |
| 14G. Copies of the consent form(s) are attached. X Yes Not applicable |
| 14H. Will this project be registered as a clinical trial? X Yes No |
| If yes, effective January 21, 2019, an informed consent form must be posted on the Federal Web site |
| after the clinical trial is closed to recruitment, and no later than 60 days after the last study visit. |
| Section 15. DEVICES & DRUGS |
| Indicate if your research includes any of the following. |
| Equipment [Researchers collecting physiological data, not testing the device] |
| (include Appendix A, the <u>Research Equipment Form</u> ) |
| Devices [Researchers planning to test devices on human subjects] |
| (include Appendix B, the <u>Device Form</u> ) |
| Materials of Human Origin |
| (include Appendix C, the <u>Biological Materials Form</u> ) |
| Drugs and Biologics |
| (include Appendix D, the <u>Drug and Chemical Usage Form</u> ) |
| MRI AT BIC To use the <u>Beckman Institute Biomedical Imaging Center</u> (BIC) in human subject's |
| research, you must obtain prior approval from the BIC (217.244.0446; <a href="mailto:ryambert@illinois.edu">ryambert@illinois.edu</a> ) and use |
| BIC-approved screening and consent forms. Attach: |
| BIC approval BIC screening form BIC consent form |
| Section 16. CONFIDENTIALITY OF DATA & PRIVACY OF PARTICIPATION |
| 16A. How is participant data, records, or specimens identified when received or collected by |
| researchers? Identifiers include, but are not limited to, name, date of birth, email address, street |
| address, phone number, audio or video recordings, and SSN. |
| No identifiers are collected |
| Direct identifiers are collected |
| Indirect identifiers (e.g. a code or pseudonym used to track participants); |
| Does the research team have access to the identity key? Yes No |
| 16B. Select all methods used to safeguard research records during storage: |
| Written consent, assent, or parental permission forms are stored separately from the data |
| Data is collected or given to research team without identifiers Data is recorded by research team without identifiers |
| Direct identifiers are removed from collected data as soon as possible |
| Direct identifiers are deleted and no identity key exists as soon as possible |
| Participant codes or pseudonyms are used on all data and the existing identity key is stored |
| separately from the data |
| Electronic data is stored in a secure, <u>UIUC-approved location</u> , please specify REDCAP and Box Health |
| VA Lieut sind data is stored in a secure, or a approved location, prease specify nebota and box field in |



| Hard-copy data is stored in a secure location on UIUC's campus, <i>please specify</i> Other, <i>please specify</i> : |
|---|
| <b>16C. How long will identifiable data be kept?</b> All identifying electronic data will be destroyed |
| immediately after data collection is completed. Audio recordings will be kept for 3 years after study |
| completion. De-identified data including COVID-19 test results will be kept indefinitely. |
| <b>16D. Describe provisions to protect the privacy interests of subjects.</b> In addition to the creation of and ongoing adherence to the DSMP and the procedures indicated earlier in this protocol, participants will be protected by a Certificate of Confidentiality issued by the NIH. Under terms of the Certificate, the researchers cannot be forced to disclose information that may identify a participant, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. However, the Certificate cannot be used to resist a demand from United States Government personnel |
| for information that is used for auditing or evaluation of federally funded projects or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). Researchers may also disclose the identity of participants who report intentions to harm themselves or others or if researchers have knowledge those participants are abusing children or elderly persons. |
| In order to further protect participants' privacy from having a navigator see their baseline information without their written consent, we will program Redcap to automatically only produce the navigation baseline report if the participant checked the yes box in the consent form. This way, navigators will only be able to see the relevant COVID-19 risk information baseline report if the participant provided written consent. |
| HIPPA protected data will be store in Redcap and Box Health. All research members with access to this information will complete a HIPPA training prior to accessing the data. Weekly staff meeting will be used to remind staff of confidentiality and HIPPA data protection protocol. |
| 16E. Describe the training and experience of all persons who will collect or have access to the data. All |
| members of the research team will complete the required CITI training and will be trained on this specific study protocol by the principal investigators. Drs. Windsor, Benoit, and Pinto have extensive experience conducting similar studies and adhere to best practices in data collection and retention. Mr. Harper, as a trained social worker and executive director of CHBC, has decades of experience in service provision, client rights and privacy, and administration of federally funded programs. Once a new research team member is hired, as part of the onboarding process at CSBH, they must complete a variety of standardized trainings on confidentiality, COVID-19, and IT security. Additionally, research team |
| members will receive training on tasks that are specific to their job expectations. Everyone will receive training on Redcap (1 hour online and homework tutorials and practices), human subjects research (CITI training), COVID-19 protocol (1 hour and ongoing training during weekly meetings), and on study protocols (includes professionalism, confidentiality, cultural humility, referral making, safety procedures). Street outreach staff will also receive training on safety while working in the field, |

confidentiality in the field, how to complete the study screener, and dos and don'ts when calling



participants (2 hours plus homework and role plays). Peer Navigators will complete an online training on Motivational Interviewing with a professional trainer (8 hours plus homework and role plays). They will also complete a 2 hour training on Navigation Services with Dr. Pinto. They will be paired with Letitia McBride, the seasoned peer navigator from New Jersey for mentorship and extra support. They will have ongoing clinical supervision weekly meetings with Dr. Windsor to review their cases, ensure fidelity, and review study protocols. The Critical Dialogue facilitator will be trained by Dr. Windsor including a period of shadowing the facilitations, role plays, and observations, until they are approved to run the sessions on their own. Finally, during staff meetings we continually identify possible training gaps and make sure these are addressed as needed. Particularly with the changes on COVID-19 recommendations, we often use the weekly meetings to review the protocol, make sure it is up to data, and that everyone has the same understanding. All of this is tracked in minutes that are recorded and saved after each meeting. This includes a table that reflects the training and the dates in which each staff completed it.

### Section 17. DISSEMINATION OF RESULTS

17A. List proposed forms of dissemination (e.g. journal articles, thesis, academic paper, conference presentation, sharing within industry, etc.).

The proposed study is purposefully planned with rapid translation, dissemination and sustainability in mind. The adaptive intervention is envisioned as an efficient and effective model that can ultimately be replicated in the field and scaled-up with high fidelity. Beginning in the research planning stage, and iteratively throughout all phases of the study, we are ensuring that the manual, once efficacious, can be disseminated among service providers across similar settings. The Collaborative Board will design a comprehensive plan to disseminate the study findings to the community at large.

Consistent with NIH policy, the PIs in the proposed application will make the data available, on appropriate terms and conditions, to the research community in a timely manner. We will follow the NIH Policy on the Dissemination of NIH-Funded Clinical Trial Information NOT-OD-16-149. The study will be registered under the Clinical Trials Registration at ClinicalTrials.gov for public posting. The study will be registered within 21 calendar days after the enrollment of the first participant, results will be submitted no later than one year after the completion of final data collection, and all required elements will be provided. Results including participant flow, demographic and baseline characteristics, outcomes and statistical analyses, adverse events, the protocol and statistical analysis plan, and administrative information will be updated on ClinicalTrials gov bi-annually (twice each study year)

| Cillical Frais.gov bi-annually (twice each study year). |
|---|
| 17B. Will any identifiers be published, shared, or otherwise disseminated? Yes No |
| If yes, does the consent form explicitly ask consent for such dissemination, or otherwise inform |
| participants that it is required in order to participate in the study? Yes |
| 17C. Do you intend to put de-identified data in a data repository? X Yes No |

| OFFICE FOR THE PROTECTION OF RESEAR | CH SUBJECTS | UNIVERSITY OF IL | LINOIS AT URBANA-C | HAMPAIGN |
|---|---|---|---|---|
| 805 West Pennsylvania Avenue, MC-095, Urbana, IL 61801 | T 217-333-2670 | irb@illinois.edu | www.irb.illinois.edu | Revised: 02/07/2020 |



If yes, explain how data will be de-identified. We will download only de-identified data from Redcap. Redcap flags any variable that contains identifiable information. We can then have the software exclude these variables automatically. The data will be exported by a doctoral student and checked by Dr. Jesus Sarol, our statistician. Moreover, the Duke data repository has additional data quality checks to make sure no identifiable information is uploaded into the system.

### Section 18. INVESTIGATOR & DEPARTMENTAL ASSURANCES

- I certify that the information provided in this application is complete and correct.
- I certify that I will follow my IRB Approved Protocol.
- I accept ultimate responsibility for the conduct of this study, the ethical performance of the project, and the protection of the rights and welfare of the human subjects who are directly or indirectly involved in this project.
- I will comply with all applicable federal, state and local laws regarding the protection of human subjects in research.
- I will ensure that the personnel performing this study are qualified and adhere to the provisions of this IRB-certified protocol.

The original signature of the PI is required before this application may be processed (electronic signatures are acceptable).

7/18/2022

Principal Investigator
Date

If the PI is not eligible to serve as PI under the Campus Administrative Manual, the applicable academic dean, institute director, or campus administrative officer indicates their approval of the researcher to act as Principal Investigator. Please note that departmental assurance only needs to be provided in the initial application.

Name of Authorizing Individual

Signature of Authorizing Individual

Date



### **Social Behavioral Research Consent Form**

TITLE OF THE STUDY: COVID-19 Treatment Cascade Optimization Study

NAME OF THE PERSONS IN CHARGE OF THE STUDY: Liliane Windsor

DEPARTMENT AND INSTITUTION: School of Social Work, University of Illinois Urbana-Champaign and

Comprehensive Behavioral Health Center

CONTACT INFORMATION: lwindsor@illinois.edu, 217-300-1782

**SPONSOR:** National Institutes of Health (NIH)

Hello, you are being asked to participate as one of 5 members of the Illinois Community Collaborative Board (ICCB). The project is being conducted by Mr. Joe Harper at the Comprehensive Behavioral Health Center and Drs. Liliane Windsor, at the School of Social Work at the University of Illinois at Urbana-Champaign, Ellen Benoit at the New Jersey Community Collaborative Board (NJCRI), and Rogério Pinto at School of Social Work at the University of Michigan.

### WHAT IS THE PURPOSE OF THIS STUDY?

The purpose of the study is to work with the ICCB to evaluate a new intervention seeking to increase testing for COVID-19 and adherence to public health recommendations in St. Clair County, IL.

### TO BE IN THIS STUDY

To be in this study you must be 18 years of age or older, live in St. Clair County, and be knowledgeable about the East St. Louis community. You must be able to speak English and willing to consent to join the study.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY?

Your participation in this study will require a two-year commitment to attend bi-monthly scheduled ICCB meetings for 2 hours each and participate in subcommittees. The ICCB will have 5 members.

### WHAT WILL HAPPEN DURING THE STUDY?

You will be asked to take an active role in the ICCB by engaging in brainstorming, planning, developing and testing the intervention. During each of the meetings, you will be asked openended questions about your thoughts on how the intervention needs to be changed, how to conduct ethical research with this vulnerable community, best practices in recruitment, implementation, data collection, and research reporting. These data will be compiled in the form of meeting minutes, video recordings, e-mail exchanges, and the research protocols. You will receive \$20 per hour of participation.

IRB Number: 22606

IRB Expiration Date: 02/27/2024

You may choose to engage in study related tasks such as recruitment and data collection. In order to protect the privacy of potential COVID-19 Optimization Study participants, we will ask you not to engage with anyone you may have a personal relationship with in any capacity as part of the study. If at any point you unexpectedly encounter someone you know in a study related activity, you will recuse yourself and notify the project coordinator and the principal investigators.

### WHAT WILL YOU DO WITH MY DATA?

All meetings are video/voice-recorded, thus agreeing to be video-recorded is a condition for participation. Recordings will be kept private in Box, a secure online cloud service. Videos will be used to aid in the development of minutes and destroyed upon minute approval (usually 2 months). Voice recording will be kept indefinitely until the ICCB decides to destroy them through a majority vote. Any ICCB member can request to listen to meeting voice recordings at any time. The recordings will be kept indefinitely to maintain a record of the research process and they may be analyzed for research purposes.

Your participation in this study will be made public through the ICCB website where your name and affiliation will be displayed as a member of the ICCB. Your name will also be published in the protocols as one of the contributors to its development.

### WHAT ARE THE POSSIBLE RISKS?

There are minimal risks associated with participation in this project. Discomfort and embarrassment are possible, but not expected. Loss of confidentiality is also a possible risk; however, several procedures will be employed to protect participants' privacy. The meetings do not require you to divulge personal, intimate, or sensitive information. You may leave the ICCB at any time by informing Dr. Windsor you no longer wish to participate.

### ARE THERE POSSIBLE BENEFITS OF THE STUDY?

You may gain personal and professional development--networking, skill building, leadership and program development, publications, research, and presentations. Since you will represent your employment organizations and/or their communities, involvement with the board may result in capacity building for those they represent. The information learned from the research project will generate empirical data which will be used by you and other researchers to guide the development of a community based intervention to combat COVID-19 and to foster future community-academic research collaborations.

### ARE THERE ALTERNATIVES TO BEING IN THIS STUDY?

Being in this study is voluntary. Choosing not to be part of the study will not result in any penalty. It will not result in any loss of benefits to you. Being in or lack of being in this study will not affect your ties with providers in the community. It will not affect your ties to the University of Illinois at Urbana-Champaign, or CBHC.

### CONFIDENTIALITY

IRB Expiration Date: 02/27/2024

Your participation in this research is public. However, all data, including meeting recordings, will be kept in Box, to which only relevant personnel will have access.

In general, we will not tell anyone any information about you. However, laws and university rules might require us to disclose information about you. For example, if required by laws or University Policy, study information which identifies you and the consent form signed by you may be seen or copied by the following people or groups: a) The university committee and office that reviews and approves research studies, the Institutional Review Board (IRB) and Office for Protection of Research Subjects; and b) University and state auditors, and Departments of the university responsible for oversight of research; and c) Federal government regulatory agencies such as the Office of Human Research Protections in the Department of Health and Human Services, and our NIH funding agency.

To help us protect your privacy, we obtained a **Certificate of Confidentiality** from the National Institutes of Health. With this Certificate, researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. We will use the Certificate of Confidentiality to resist any demands for information that would identify you, with the following exceptions:

- 1) The certificate cannot be used to resist a demand for information from personnel of the agency sponsoring the project and that will be used for auditing or program evaluation of agency-funded projects.
- 2) You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research.
- 3) If you give another person or organization your written permission to receive research information, then we may not use the Certificate to withhold that information.

### PAYMENT FOR BEING IN THE STUDY

You will receive \$20 per hour of meeting participation.

### **LEGAL RIGHTS**

You will not lose any of your legal rights by submitting this consent form.

### **CONTACT INFORMATION**

If you have questions or suggestions about the study or the procedures, you may contact Dr. Liliane Windsor at (217) 300-1782 (lwindsor@illinois.edu). If you have questions about your rights as a research subject, including concerns, complaints, or to offer input, you may call the Office for the Protection of Research Subjects (OPRS) at 217-333-2670 or e-mail OPRS at irb@illinois.edu. You may if you would like to complete a brief survey to provide OPRS feedback about your experiences as a research participant. Please follow the link here or through a link on the OPRS website: https://oprs.research.illinois.edu/. You will have the option to give feedback without using your name. You have the option to talk about your concerns without



IRB Number: 22606

IRB Approval Date: 02/28/2023 IRB Expiration Date: 02/27/2024

using your name. You may provide your name and contact information for follow-up purposes. You will receive a copy of this information in your email. Feel free to download a copy using the link below for your records.

If you choose to participate, please print and sign your name and date on the lines below.

| Participant Name (print): |
|-------------------------------|
| Participant Name (signature): |
| Date: |

IRB Approval Date: 02/28/2023 IRB Expiration Date: 02/27/2024



### **Social Behavioral Research Consent Form**

TITLE OF THE STUDY: COVID-19 Treatment Cascade Optimization Study

NAME OF THE PERSONS IN CHARGE OF THE STUDY: Liliane Windsor

**DEPARTMENT AND INSTITUTION:** School of Social Work, University of Illinois Urbana-

Champaign and Comprehensive Behavioral Health Center

CONTACT INFORMATION: lwindsor@illinois.edu, 217-300-1782

**SPONSOR:** National Institutes of Health (NIH)

You are being asked to join a voluntary research study. There are study goals. One goal is to develop a way to increase COVID-19 testing. Another goal is to encourage people to do things like wear masks and practice social distancing to avoid COVID-19. This study checks how the three different interventions work for people. People are put into to a group by chance. Your group may meet for six months, or it may be done meeting after one survey. You may be asked to fill out 1 to 5 surveys. You may be asked to go to one group meeting. We may call you one to two times to answer questions on the phone. There are some risks to entering this study: 1) We ask private questions about medications you are taking, disabilities, if you currently use drugs, whether you have any illness that makes you at risk to develop severed COVID-19 symptoms; 2) There is a small chance that people could find out what your answers were. 2) You may feel some strong feelings answering the questions including feeling sad. There are no direct benefits to join this study. You do not have to agree to join the study.

### WHAT IS THE PURPOSE OF THIS FORM?

This form will help you decide if you want to join this study. This form describes the purpose, procedures, benefits, risks, discomforts, and protections of the study. It describes different options that are available to you. It also describes your right to quit the study at any time. Please ask as many questions as you like to fully understand the study. After you know about the study please decide if you would like to join. You will be asked if you agree to take part in it. You can download a copy of this consent form. The form is in the e-mail invitation you received. You may show this consent form to family. You may show it to other doctors and medical staff. Not only that, but you may show this form to your friends. You may want to talk about it with them before you sign the form. They may help you decide if you want to be part of the study. This study is funded by the National Institute of Allergy and Infectious Disease (NIAID). It is part of the National Institutes of Health (NIH) in Washington, DC. The Principal Investigators are Liliane C. Windsor of the University of Illinois at Urbana-Champaign, Ellen Benoit of NJCRI, Joe Harper of CBHC, and Rogério Pinto of The University of Michigan. The NIH is part of the United States Department of Health and Human Services. The NIH's purpose is to find new information that will lead to better health for everyone. This study is part of the RADx-UP program. The NIH funded (gave money to) the RADx-UP program. RADx-UP stands for Rapid Acceleration in Diagnostics (in) Underserved Populations. RADx-UP is a health research program to learn more about COVID-19 disease. If you join RADx-UP, we will gather some data (information) about you. We will send the data to The Duke Clinical Research Institute (DCRI). This research group was chosen by the National Institute of Health (NIH). They will combine the data collected from everyone taking part in RADx-UP studies. Your data will be added together with other people's data who join RADx-UP. Researchers will study the RADx-UP data. They will use this data to try to help people who are at risk for or with COVID-19.

IRB Expiration Date: 02/27/2024

You are being asked to be in this study because you told us that you may be at high risk of getting COVID-19 or experiencing problems from it.

### TO BE IN THIS STUDY

To be in this study you must be 18 years of age or older. You must be either at high risk of contracting COVID-19 or developing problems from it. You must be able and willing to consent to join the study.

## HOW LONG THE STUDY WILL LAST AND HOW MANY PEOPLE WILL BE IN THE STUDY?

During this study you may be asked to complete 1 to 5 research interviews. The interviews may last between 5 minutes and 60 minutes. You may have to attend one group meeting. The group meetings are about 1 hour. There may be two 15 to 30-minute phone calls or in-person sessions. Some people will complete the study after the first interview. It may take about 6 months to complete the meetings and all the interviews. You may be asked to be interviewed online. The interview might be over the phone. The interview if safe, might be in person. Different people will be picked by chance to do different activities. We expect to recruit a total of 1218 people to be in this study. All participants will be adults. They may be high risk of being exposed to the COVID-19 virus. They may be high risk of developing health issues from a COVID-19 infection. They may be both.

### WHAT WILL HAPPEN DURING THE STUDY?

If you agree to join the study, we will ask you to take a COVID-19 test at CBHC. We may ask you to attend a session(s) with a peer navigator or a licensed clinician. These sessions could last up to 30 minutes. The sessions may be on the phone or in-person. The number of sessions will depend upon your version of the program. You will not be able to choose which group you will be joining. This means you will be in a group by chance. The groups include a peer navigation group, an informational brochure group, a brief individual counseling group, or a group intervention called Critical Dialogue. Critical dialogue meets once for an hour. The study will take 6 months, no matter which group you join. We may also ask you to complete one to 5 online surveys. The surveys are called baseline, follow-up 1, 2, 3, and 4. We will ask to get your results from the COVID-19 test you take at CBHC.

Some questions in the surveys will ask you for information about yourself. Examples include gender, race, ethnicity. The survey will ask about your health and living situation. The survey will ask about vaccines, and COVID-19. The survey will include questions about what you went through during the pandemic. The COVID-19 test will have a sample taken from the inside of your nose with a swab. You may do the swab yourself. You may have a member of the clinical study team do it. The sample will be analyzed by a machine at CBHC. The results should be available within 20 minutes. A staff member will tell you your results in private. If your results are positive, you will receive information on how to quarantine. You will also get information on medical care. If your results are negative, you will receive information on how to stay safe. The information will include how to avoid infection. The navigation group, will have a peer navigator. The peer navigator be able to see the information you shared in the first survey. The peer navigator will call you to talk about your COVID-19 risk. 3

IRB Expiration Date: 02/27/2024

Thirty five participants will be selected to complete a phone interview. The phone interview will be about 30 minutes. The interview will be about their experience with the study. It will include their feelings about COVID-19 testing. It will also include their feeling about public health safety measures. The information you give us will be kept private. The information will include results from the COVID-19 test. Your answers to the questions in this study will be completely confidential. If you do not want to answer a question, you may refuse to answer it. You may refuse to participate in a certain part of the study. If you refuse, there will not be a penalty. You may receive a COVID-19 swab test without joining the study.

### WILL HEALTH INFORMATION ABOUT YOU BE CREATED, USED OR SHARED WITH OTHERS DURING THIS STUDY?

Researchers are required to protect your health information. Your health information is protected by state and federal laws. It is protected by the Health Insurance Portability and Accountability Act (HIPAA). This form tells you how the researchers in this study may use your health information. It tells you how it may be shared. By signing this form, you are letting Dr. Windsor (head researcher) and the research team to obtain, use, store, and share protected health information that identifies you for the purposes of this research. The health information is specific to your COVID-19 test results. These results will be collected at the Comprehensive Behavioral Health Center (CBHC). During this study, the researchers may use or share your COVID-19 test results with:

- Each other and with other researchers involved with the study.
- With the National Institutes of Health (NIH). This is required to conduct the research. It is required to confirm the results of the research.
- With members of the University committee and office, the Institutional Review Board (IRB) and the Office for the Protection of Research Subjects. They review and approve research studies.
- With other government representatives and University employees. They are responsible for ethical, governing, or financial supervision of research.

Once the study ends, all information that identifies you will be removed. This is called de-identified information. Then this form will no longer apply. If it is allowed by law, your information may be given and used by others. It might be used for other purposes, such as other research projects. While you are taking part in this research, you will receive your COVID-19 test results. In an emergency, the research team can give your results to your doctor.

How will your health information be protected?

The researchers and the NIH agree to protect your health information. They will only share this information as described above. The agencies listed above may not be required to protect it. If it is allowed by law, they may share your information with others. They may do this without your permission.

Your permission to share your health information in this form will end at the end of the study. You may change your mind at any time. To end your permission, send an e-mail to Dr. Liliane Windsor at lwindsor@illinois.edu. If you cancel this permission, you may not be allowed to take part in the study. The researchers will delete your COVID-19 test results from the study.

IRB Expiration Date: 02/27/2024

### Right to Refuse to Sign this Authorization

You do not have to sign this consent/permission form. Not signing this form will not affect your ability to receive treatment. It will not affect your ability to make payments. It will not affect your ability to enroll in any health plans. It will not affect your eligibility for other medical benefits. If you have questions or concerns regarding your privacy rights under HIPAA, you should contact the University of Illinois HIPAA Privacy Office. Their phone number is (844) 341-2201. Their email is hipaa@uillinois.edu.

By clicking the agree button below, you are providing permission. This permission is for the researcher to gather your COVID-19 test results. This permission includes the uses of your test results. This permission is to share your test results. All the of the test results are used for the purposes of this research.

| ı | agr | ee | |
|---|-----|-----|-------|
| ı | do | not | agree |

### WHAT WILL YOU DO WITH MY DATA?

Our research team and the Duke Clinical Research Institute (DCRI) will keep your data confidential. This means they will take extra precautions to make sure no one sees your information without your consent. The data from other people who are in the RADx-UP program will also be confidential. Researchers will use the data to learn more about COVID-19. The researchers will also use the data to learn about other diseases and conditions. The DCRI will build two RADx-UP databases. Databases are systems that hold electronic information. The first database will only hold information that can identify you. This data is called identifiable information. Examples of the data are your name, address, email, and gender.

- This data will be kept at the DCRI. The DCRI will not share this data with the NIH.
- Only if you agree, the DCRI will keep this information. To show you agree please click the box below. This will allow us to contact you for future research studies. If you do not agree, this information will only stay with your study team.
- The data will stay in a password-protected secure electronic system. Only staff at DCRI will be able to see this information. They are in charge of maintaining the security of your data.
  - The second database will not hold information that identifies you. It will hold all the other information you agree to give.
- You will be assigned a study code. You will only be identified in this database by this study code.
- It will not contain your name. It will not include other identity information.
- We plan to keep this non-identifiable data in a secure database for COVID-19 research.
   We plan to transfer it to the NIH. Other researchers may use this data in other studies.
   These researchers are not on this consent form.

IRB Expiration Date: 02/27/2024

• When using this data, researchers will only have access to your non-identifiable data. Researchers cannot link the data back to you.

• When we share this data, we will not contact you. We will not ask your permission. This is because the data cannot be linked back to you.

Please select the permissions you are willing to give DCRI:

| I agree to let the DCRI collect only my ZIP code. I agree to collect the other information as ted above. |
|---|
| I agree to let DCRI contact me for future research as stated above. |

### WHAT ARE THE POSSIBLE RISKS?

There are risks in this study. One risk is an accidental loss of private information. Another risk is potential emotional discomfort. We will ask you questions about medications you are taking, disabilities, if you currently use drugs, whether you have any illness that puts you at risk to develop severed COVID-19 symptoms. The prospect of testing positive for COVID-19 may cause fear and anxiety. Receiving a positive COVID-19 test result can be upsetting. Some people may find the content of intervention sessions disturbing.

We will take many steps to protect your identity. We will take many steps to keep your responses private (see details below). There is a small chance that confidentiality may be lost. You may participate in the Critical Dialogue group discussion. Peers in your group will learn information about you that you choose to share. We will ask everyone in the Critical Dialogue group to respect the privacy of others. We will ask them to treat anything said in the group as confidential. Please remember other participants may not follow this request. It is possible that data could be stolen if our server is hacked. We will take every precaution to prevent this from happening. We will use locked files. We will have password-protected secured servers to keep your information safe. Researchers are required to report child abuse. They are required to report people who are in immediate danger. The researcher will notify the correct authorities. If you begin to talk about this during an interview, it will not be kept a secret. The researcher will stop you and tell you that such information cannot be kept a secret.

### ARE THERE POSSIBLE BENEFITS OF THE STUDY?

We cannot guarantee that being in this study will have positive effects. We hope that this study will be helpful to you. We hope it will help members of your community. The positive effect includes detecting, treating, and preventing the spread of COVID-19 cases. We also hope that participants will benefit from referrals. These referrals are resources to housing, food, and other basic needs that help maintain health. If participants express a need for mental health assistance at any time, the project team can either make referrals.

### ARE THERE ALTERNATIVES TO BEING IN THIS STUDY?

IRB Expiration Date: 02/27/2024

Being in this study is voluntary. Choosing not to be part of the study will not result in any penalty. It will not result in any loss of benefits to you. Being in or lack of being in this study will not affect your ties with providers in the community. It will not affect your ties to the University of Illinois at Urbana-Champaign, or CBHC.

### WILL IT COST ANYTHING TO BE IN THIS STUDY?

There will be no cost to you for being in the study.

### **CONFIDENTIALITY**

We will make sure that your privacy and confidentiality are protected. Will not let your name appear on any research records or results. We may ask you for contact information. This will be your phone number and address. We ask this, so we can reach you to schedule follow-up interviews. Contact information may be kept in the project manager's locked filing cabinet. Contact information may be kept in a password-protected file. There will be a code number placed on all the interview documents. There will be a code number on all test results. You will use a code name during interviews and in group sessions. Your code number to your name is only available to trained research team members with permission. Your comments will be kept confidential. Only the study's researchers will have access to your information. They will use it to schedule appointments. Things that you say throughout the study will be written down. It will be written in ways that will protect your identity. Specific things you say, will never refer to you by name or number. For example, we might report that during one group session, "four people tested positive for COVID-19."

Once the study is completed, other researchers may ask to use the data. Sharing data is an important way to help other studies. We will make the data available to others, but only if we believe your identity and privacy are protected. To share the data, we will require an agreement that has the following conditions: (1) a commitment to use the data only for research purposes and not to identify any individual participant; (2) a commitment to protect the data using appropriate tools and computer technology; and (3) a commitment to destroy or return the data after analyses are completed. We will remove all personal identifiers from the data before we will allow it to be used by other researchers.

To help us protect your privacy, we obtained a Certificate of Confidentiality from the National Institutes of Health. This Certificate states, researchers cannot be forced to disclose information that may identify you, even by a court subpoena, in any federal, state, or local civil, criminal, administrative, legislative, or other proceedings. We will use the Certificate of Confidentiality to resist any demands for information that would identify you, with the following exceptions:

- 1) The certificate cannot be used to resist a demand for information from NIH personnel and that will be used for auditing or program evaluation of agency-funded projects.
- You should understand that a Certificate of Confidentiality does not prevent you or a member of your family from voluntarily releasing information about yourself or your involvement in this research.

IRB Expiration Date: 02/27/2024

3) If you give another person or organization your written permission to receive research information, then we may not use the Certificate to withhold that information.

4) Mandated reporting of ongoing child abuse or immediate danger.

All project staff will be trained in how to protect your data. They will sign a pledge of confidentiality. Privacy will be protected when contacting participants about joining the study and participation. Only study staff will talk with you directly. The other staff may leave a message if you ask. In general, we will not tell anyone any information about you. When this study is discussed or published, no one will know that you were in the study. Faculty, staff, students, and others with permission or authority to see your study information will maintain its privacy. They will do this to the extent permitted and required by laws and university policies.

### PAYMENT FOR BEING IN THE STUDY

You will receive compensation for each interview or critical dialogue activity you join. This includes \$30 for the baseline interview. It will also include \$40 for each follow-up interview you complete. You will also receive \$30 for attending the critical dialogue session. You might be selected by chance for an in-depth individual interview. If you complete that interview, you will receive an additional \$50. You may receive a minimum of \$30 and a maximum of \$270. To receive it, you must be eligible to participate in all possible research interviews. You must complete all the interviews during the 6 months.

### **LEGAL RIGHTS**

You will not lose any of your legal rights by submitting this consent form.

### **CONTACT INFORMATION**

If you have questions or suggestions about the study or the procedures, you may contact Dr. Liliane Windsor at (217) 300-1782 (lwindsor@illinois.edu). If you have questions about your rights as a research subject, including concerns, complaints, or to offer input, you may call the Office for the Protection of Research Subjects (OPRS) at 217-333-2670 or e-mail OPRS at irb@illinois.edu. You may if you would like to complete a brief survey to provide OPRS feedback about your experiences as a research participant. Please follow the link here or through a link on the OPRS website: https://oprs.research.illinois.edu/. You will have the option to give feedback without using your name. You have the option to talk about your concerns without using your name. You may provide your name and contact information for follow-up purposes. You will receive a copy of this information in your email. Feel free to download a copy using the link below for your records.

### AGREEMENT TO BE IN THE STUDY

I have read this entire form and I understand it completely. All of my questions regarding this form have been answered to my satisfaction. All my questions about this study have been answered to my satisfaction. I understand that my participation in this research project is voluntary. I know that I may quit the study at any time. Quitting will not harm my future medical care. It will not cause any loss of benefits to which I might be entitled. I know the researcher



IRB Number: 22606

IRB Approval Date: 02/28/2023 IRB Expiration Date: 02/27/2024

may decide that I should no longer be in this study. I know this may happen at any time. I agree to receive testing and medical services from CBHC. I agree to have my information added to the electronic medical records.

| added to the electronic medical records. |
|---|
| Yes No By clicking the Yes button below, I am agreeing to participate in this study. I understand that I have not waived any of my legal rights. |
| Yes<br>No |
| I understand that I may be in the Navigation Services group. My peer navigator will look at my COVID-19 risks answers in the baseline survey. My peer navigator will keep my answers confidential. It will be used to make my navigation session relevant to my needs. |
| Yes<br>No |
| CONTACT FOR FUTURE STUDIES |
| The CBHC and the University of Illinois have health-related studies. They seek research participants. We have a study participant bank. Would you like us to add your name and contact information to it? If you note yes, we may invite you to join studies. |
| Please check your choice: |
| I consent to the study staff adding my information to study bank. I am not interested in being contacted about future studies. |